CLINICAL TRIAL: NCT02989428
Title: Cardiovascular Health in Patients With Primary Hyperparathyroidism: Effect of Parathyroidectomy on Cardiovascular Health: A Randomized Controlled Trial
Brief Title: Effect of Parathyroidectomy on Cardiovascular Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UAarhus170879
Record Dates: First submitted 2016-12-02; First posted 2016-12-12 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2018-04

CONDITIONS: Primary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Primary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early parathyroidectomy group (Experimental): Parathyroidectomy (surgery), is performed as soon as possible in the experimental group after randomization.
  Interventions: Procedure: Early parathyroidectomy group (EPTX-group)
- Late parathyroidectomy group (No Intervention): Parathyroidectomy (surgery), is performed three months after study inclusion.

INTERVENTIONS:
Procedure: Early parathyroidectomy group (EPTX-group) — Participants will undergo parathyroidectomy as soon as possible
  Arms: Early parathyroidectomy group

SUMMARY:
The aim of this study is to establish whether patients with mild primary hyperparathyroidism (PHPT) have an increased risk of cardiovascular diseases. The primary outcome is to determine whether arterial stiffness and blood pressure will decrease in patients with mild PHPT 3-month after parathyroidectomy (PTX).

DETAILED DESCRIPTION:
Background:

The cardiovascular manifestation of primary hyperparathyroidism (PHPT) has been debated in many years. PHPT was once a highly symptomatic disease with severe symptoms. Today, the clinical presentation of the disease is often asymptomatic or with few symptoms at diagnose. This may be the reason why the literature regarding this area is conflicting. Studies have observed an increased mortality cause by cardiovascular diseases (CVD) in moderate to severe disease, whereas other studies with focus on mild disease observed no increased risk of mortality. A shift in the clinical presentation of the disorder to a more asymptomatic appearance makes it pivotal to investigate CVD risk in patients with PHPT before and after surgery. Large-arterial stiffness is known to be a predictor of cardiovascular events and all-cause mortality. Measurement of carotid-femoral pulse wave velocity (PWV) is considered as the gold standard for non-invasive measurement of arterial stiffness. To date, only few studies have investigated the relationship between PWV and PHPT. In three prospective studies the authors reported a significant increase in PWV preoperative in PHPT patients compared to controls. 6-month after parathyroidectomy two of the studies observed a significant decrease in PWV, where one study observed a non-significant decrease. Another study by Ring et al observed only a slightly, but significant increased PWV in PHPT patients compared to controls and no changes after surgery at 1-year follow-up. However, a study by Tordjman et al observed no differences in PWV among PHPT patients compared to controls. In addition, other studies have explored the relationships between arterial stiffness and PHPT using either augmentation index (AIx) or carotid intima-media thickness (IMT) as predictors for arterial stiffness. Three studies with focus on AIx reported an increased AIx in PHPT patients, whereas two other studies observed no increased AIx in PHPT patients compared to controls. Using the IMT methods, two studies reported a significant increased IMT in PHPT patient preoperative compared to controls and a significant decrease after parathyroidectomy. Furthermore, a study by Walker et al observed an increased IMT in PHPT patients compared to controls but in a subsequent follow-up study there was no changes in IMT after surgery. In contrast, one study reported no differences in IMT in PTHP patients before and after surgery. Most research so far has focussed on different methods for measurements of arterial stiffness which makes a comparison among studies difficult. More research with focus on one of the methods is necessary.

Another clinical aspect of PHPT is the increased prevalence of hypertension compared to the general population. Previous research findings into parathyroidectomy's effect on hypertension have been inconsistent and contradictory. Four studies reported no effect of parathyroidectomy on preoperative hypertensive patients and in two studies they observed an increased incidence in hypertension after surgery. However, in four other studies they observed a significant postoperative reduction in systolic and diastolic BP among known hypertensive patients at follow-up.

Nevertheless, much uncertainty still exists and more research investigating the relationship between BP and arterial stiffness pre- and postoperative is required. PWV is considered the gold standard for non-invasive measurements of arterial stiffness and a predictor for cardiovascular events and all-cause mortality. It is therefore the best approach to assess the association of PHPT and cardiovascular risk in combination with BP. In addition, until now study design has been prospective with small population sizes. Therefore, we need to perform a randomized controlled trial (RCT) comparing arterial stiffness and blood pressure (BP) in patients with mild PHPT pre- and post-operative. This study will be the first performed randomized controlled trial (RCT) investigating arterial stiffness and BP in patients with PHPT. Hopefully, this study will be able to establish the cardiovascular risk in patients with mild PHPT and have an influence on future international guidelines for management of PHPT.

Aim:

The aim of this study is to establish whether patients with mild PHPT have an increased risk of cardiovascular diseases. The primary outcome is to determine whether arterial stiffness and BP will decrease in patients with mild PHPT 3-month after parathyroidectomy (PTX). Arterial stiffness will be assessed as PWV and BP as sitting- and 24-hour BP. In addition, the study will evaluate the effect of PTX on serum cholesterol and other markers of cardiovascular risk.

Hypothesis:

1. Patients with PHPT have an increased cardiovascular risk assessed by BP, PP (central pulse pressure) and arterial stiffness.
2. PWV, PP and BP in patients with PHPT will decrease 3-month after PTX.

Study design:

The study will be performed as a RCT enrolling patients with PHPT. Participants will be assessed at baseline and subsequently randomized to one of two study groups, i.e., a group in which PTX is performed as soon as possible ("early PTX group" [EPTX-group]) and a group in which PTX is performed three months after study inclusion ("late PTX group" [LPTX-group]). Follow-up will be performed 3 months after PTX in the EPTX-group and after 3 months of observation in the LPTX-group. All enrolled participants will undergo PWV, PP, BP and blood samples at baseline and at 3-month follow-up. Since women are affected by the disease substantially more often than men are, the randomization will be performed as a bloc randomization with 4 participants in each bloc. In each bloc two participants will be randomized to either EPTX or LPTX. With a minimum of 80 participants (see statistic section for power calculation) enrolling in the study 20 blocs will be created. Four of the blocs will be allocated to the men in the study. The first man included will start with the randomization number 64 and then the following men will be given numbers up to 80. If the men included in the study are an unequal number, a bloc with a mix of women and men will be constructed. Because of the inclusion criteria in the intention to treat analysis (see below) more than 80 people will be included to calculate for drop outs. The same principle for bloc randomization as describe above will be followed creating additional blocs with four participants in each. If more than 16 men are included they will continue receiving numbers from 81. For the likelihood to demonstrate an effect of PTX on the cardiovascular risk in PHPT patients, the analysis will be restricted only to the population that obtain a normal p-calcium after PTX.

Aarhus University Hospital is the primary center for diagnostic and treatment of PHPT in the Region of Central Denmark. Hence, all referred patients with possible PHPT will be contacted during their hospital visit. Participants fulfilling the diagnostic criteria for PHPT will be asked for participation in the project.

PHPT is defined as elevated p-calcium of minimum 3 measurements and parathyroid hormone in the upper one-third of or above the reference range.

Measurements:

Questionnaires: Height and weight will be measured on all participants. Additional information about each participant will be collected through interview/questionnaires which concerns: previous and current diseases, history of fractures, smoking status, consumption of alcohol and use of medications. Medications covers all prescribed medication, calcium and vitamin-D supplementation and natural medicine. Regarding females we will collect information about age at menarche, pregnancy, labour, menopause, and previous and current use of hormonal contraceptives.

For assessment of quality of life all participants will be asked to fill out 36-Item Short Form Survey (SF-36) either in written form or online at baseline and at 3-month follow-up.

Blood pressure: After 5 minutes of rest in sitting position BP will be measured in both right and left upper arm. Recorded BP will be measured in the arm with the lowest BP with three following measurement performed with 2 minutes rest in between. The average of the last 2 measurement will be recorded. Furthermore, a 24-hour BP measurement will be performed on each participant in the non-dominant arm.

Tonometry: In a supine position after 10 minutes of rest PP and PWV are assessed using the SphygmoCor system (AtCor Medical, cuff-based system) with applanation tonometry. The test will be performed on fasting participants in the morning both at baseline and at follow up to avoid diurnal variation. A cuff is placed around right thigh while measurements will be performed on the right carotid arterial. The carotid-femoral PWV is estimated as the distance traveled divided by transit time. A minimum of 2 readings are performed and where there is more than 0.5 m/s difference in the two measurements a three one is performed.

Biochemistry: Blood samples will be collected in the morning fasting, through a venepuncture, at baseline and at 3-month follow-up. The concentrations of albumin, total and ionized calcium, creatinine, hbA1C, total cholesterol, LDL, HDL, triglycerides, P-PTH, P-25(OH)D will subsequent be determine. Plasma will be frozen down for later analysis of apolipoprotein (Apo-A and Apo-B), high-sensitive CRP, interleukin-6, TNF-alfa, VCAM-1, fibrinogen, von Willebrand factor and CD40L.

Statistic:

The difference between the two groups will be assessed using either a paired t-test or Mann-Whitney U-test depending on distribution for continuous variables. Pearson's correlations coefficient will be used to determine relationships between variables. Multiple-linear regression analysis with PWV, PP and BT as the dependents variables will be performed adjusting for age, BP, height, smoking status, BMI, anti-hypertensive medications and hyperlipidaemia. With a sample size of 40 participants in each group the study has an 84 % power to detect a significant difference in PWV of 1 m/s between treatment and control groups. This is under the assumptions that a healthy person have a mean PWV of 8.4 m/s and a standard deviation of 1.5 m/s. Assuming a mean arterial blood pressure of 91 (±8) mm Hg, a sample size of 40 participants in each group will allow for a 80 % statistical power to detect a between group difference of 5 mm Hg (p<0.05).

Since the analysis only will be restricted to the participants in the EPTX group obtaining normal p-calcium, we will aim to recruit 80-100 participants.

Ethical aspects:

The study is performed under the current guidelines developed in the Helsinki-declaration concerning research with humans. Participants will be informed orally and in written about the project's aim, execution and possible side effects. The project is entirely voluntarily and the participants can withdraw their consent anytime during the study, without any reasons. It will not affect their ongoing and future treatments if a participants decide to withdraw. Only participants given full consent orally and in written will be enrolled in the study.

The waiting period for a PTX operation at the Aarhus University Hospital is normally 2-3 month and therefore the enrolled participants in the control group will maximum wait an extra 2-4 week. As PHPT most often is a disease which develops over several years, postponement of the treatment by surgery for a few weeks in the LPTX-group is not presumed to carry any risk for the participants.

ELIGIBILITY:
Inclusion Criteria:

* Primary hyperparathyroidism
* Referred to Aarhus University Hospital with the diagnose; primary hyperparathyroidism
* Participant is over 18 years old, able to understand and sign consent form

Exclusion Criteria:

* Familial hypocalciuric hypercalcaemia
* Multiple endocrine neoplasia (MEN)
* Parathyroid cancer
* Renal disease - GFR < 60 ml/min
* Major heart surgery
* Known coronary heart disease
* NYHA III-IV
* Known with pacemaker
* Arrhythmia e.g. atrial fibrillations or flutter, Second- and third-degree atrioventricular block, sinoatrial depolarization of < 40 or > 160 beats per minute.
* Ongoing treatment with beta-blockers
* Severe manifest osteoporosis with multiple fractures
* Severe hypercalcemia: p-ionised calcium > 1.70 mmol/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Decrease in arterial stiffness after parathyroidectomy | 3 month
  Decrease in arterial stiffness measured by pulse wave velocity 3 month after parathyroidectomy

SECONDARY OUTCOMES:
Decrease in systolic blood pressure after parathyroidectomy | 3 month
  Decrease in systolic blood pressure after parathyroidectomy measured by 24-hour blood pressure monitoring
Decrease in diastolic blood pressure after parathyroidectomy | 3 month
  Decrease in diastolic blood pressure after parathyroidectomy measured by 24-hour blood pressure monitoring
Decrease in central pulse pressure after parathyroidectomy | 3 month
  Decrease in central pulse pressure after parathyroidectomy measured by pulse wave analysis
Decrease in systolic blood pressure after parathyroidectomy | 3 month
  Decrease in systolic blood pressure after parathyroidectomy measured by ambulatory blood pressure
Decrease in diastolic blood pressure after parathyroidectomy | 3 month
  Decrease in diastolic blood pressure after parathyroidectomy measured by ambulatory blood pressure

OTHER OUTCOMES:
Quality of Life (QoL) | 3 month
  SF-36 questionnaire version 2

CONTACTS AND LOCATIONS:
Overall Officials: Lars Rejnmark, M.D, PhD, Principal Investigator — Department of Endocrinology and Internal Medicine
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ejlsmark-Svensson H, Rolighed L, Rejnmark L. Effect of Parathyroidectomy on Cardiovascular Risk Factors in Primary Hyperparathyroidism: A Randomized Clinical Trial. J Clin Endocrinol Metab. 2019 Aug 1;104(8):3223-3232. doi: 10.1210/jc.2018-02456. PMID 30860588